CLINICAL TRIAL: NCT00562653
Title: Study of Autoantibodies in Infective Endocarditis
Brief Title: Autoantibodies and Clinical Symptoms in Infective Endocarditis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Ministry of Health, Israel (Other Government)
Other Study IDs: sourasky medical centrs
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Infective Endocarditis
Keywords: profile autoantibodies; clinical symptoms
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: infective endocarditis patients before treatment
- 2: infective endocarditis treatment after treatment
- 3: control

SUMMARY:
The purpose is to evaluate autoantibodies in infective endocarditis patients before, at the beginning of treatment, and after the end of the treatment, and to correlate the autoantibodies in the presence of clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Infective endocarditis patients by DUKES criteria

Exclusion Criteria:

* HIV positive
* Patients suffering from other infective diseases other than endocarditis.
* Patient suffering from collagen diseases for example: systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), mixed connective tissue disease, and scleroderma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: infective endocarditis patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Study Completion 2008-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bogusllavsky, MD, Principal Investigator — Sourasky Medical Center, Internal Medicine
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel